CLINICAL TRIAL: NCT06104696
Title: Comprehensive Geriatric Assessment in Kidney Transplantation
Acronym: CoGeriaTx
Status: Recruiting | Type: Observational
Sponsor: Institute for Clinical and Experimental Medicine (Other Government)
Responsible Party: Principal Investigator, Silvie Rajnochova Bloudickova, Head of Outpatient Clinic of Deparment of Nephrology, Transplant Center, Institute for Clinical and Experimental Medicine
Other Study IDs: Geriatrics
Record Dates: First submitted 2023-08-04; First posted 2023-10-27 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Kidney Transplant; Complications; Frailty Syndrome; Depressive Syndrome
Keywords: kidney transplantation; geriatric; frailty; depression; pretransplant evaluation; comprehensive geriatric assessment; posttransplant
MeSH Terms: conditions — Frailty; Depressive Disorder; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood and urine samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Non-frail: Group of patients which will meet the criteria for non-frail according to the result of functional examination.
  Interventions: Procedure: Functional geriatric assessment
- Pre-frail: Group of patients which will meet the criteria for pre-frail according to the result of functional examination.
  Interventions: Procedure: Functional geriatric assessment
- Frail: Group of patients which will meet the criteria for frail according to the result of functional examination.
  Interventions: Procedure: Functional geriatric assessment

INTERVENTIONS:
Procedure: Functional geriatric assessment — Examination of physical and mental status using standardized tests.

SUMMARY:
This observational study aims to analyze the results of comprehensive geriatric assessment and to monitor the development of functional status in geriatric kidney transplant candidates and recipients.

DETAILED DESCRIPTION:
Kidney transplantation represents the best therapeutical option in patients in end stage kidney disease. At present, increasing number of older patients are referred for kidney transplantation. Patients' functional status has been shown to be associated with transplant outcomes.

The comprehensive geriatric assessment (CGA) of functional and mental status in older kidney transplant candidates might play an important and supportive role in the pre-transplant evaluation process, including acceptance for transplantation. In kidney transplant recipients, this examination might be useful to evaluate the impact of pre-transplant status on post-transplant course. Also in KTR, CGA may contribute to the improvement of functional status and quality of life independently from the graft function.

ELIGIBILITY:
Inclusion Criteria:

* kidney transplant candidates aged 60+ years
* kidney transplant recipients aged 60+ years

Exclusion Criteria:

* kidney transplant candidates aged below 60 years
* kidney transplant recipients aged below 60 years

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Kidney transplant candidates and kidney transplant recipients aged 60+ years.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-01-02 (Actual); Primary Completion 2025-01-02 (Estimated); Study Completion 2040-01-02 (Estimated)

PRIMARY OUTCOMES:
Frailty syndrome (Fried frailty phenotype) | 2020-2040
  Geriatric assessment of frailty syndrome in kidney transplant candidates and recipients. Evaluation of frailty syndrome based on Fried frailty phenotype, Short Physical Performance Battery (SPPB) and complex comprehensive geriatric assessment including cognitive frailty (Montreal Cognitive Assessment MoCA).
Acceptance for kidney transplantation (Number of patients listed for kidney transplantation and number of transplanted patients) | 2020-2040
  Acceptance for kidney transplantation based on both geriatric and nephrologic evaluation. Number of patients listed for kidney transplantation,number of transplanted patients and number of patients not accepted for transplantation.
Outcomes of kidney transplantation (Graft and patient surival, number of patients with related adverse events) | 2020-2040
  Outcomes of kidney transplantation based on both geriatric and nephrologic evaluation.
  Short- and long-term patient and graft survival, graft function, post-transplant related adverse events (infection rate, MACE, death, days of hospitalisation).
Functional status evaluated by comprehensive geriatric assessment | 2020-2040
  Functional status evaluated by comprehensive geriatric assessment in geriatric kidney transplant candidates and recipients including evaluation of mobility (Short Physical Performance Battery, SPPB, walking speed m/s, muscle strenght measured by hand-grip) and cognition (Montreal Cognitive Assessment, MoCA), self-sufficiency and/or dysability (Activities of Daily Living, ADL, Instrumental Activities of Daily Living, IADL).
Depressive syndrome (amount of depressive symptoms measured by GDS scale) | 2020-2040
  Depressive syndrome in geriatric kidney transplant candidates and recipients. amount of depressive symptoms measured by GDS (Geriatric Depression Scale) scale by Yesavage.

CONTACTS AND LOCATIONS:
Overall Officials: Silvie Rajnochova Bloudickova, MD,PhD, Study Director — Department of Nephrology, Institute for Clinical and Experimental Medicine; Hana Vankova, MD,PhD, Principal Investigator — Charles University, Czech Republic
Locations (1):
- Department of Nephrology Transplant Centre IKEM, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Result] Kobashigawa J, Dadhania D, Bhorade S, Adey D, Berger J, Bhat G, Budev M, Duarte-Rojo A, Dunn M, Hall S, Harhay MN, Johansen KL, Joseph S, Kennedy CC, Kransdorf E, Lentine KL, Lynch RJ, McAdams-DeMarco M, Nagai S, Olymbios M, Patel J, Pinney S, Schaenman J, Segev DL, Shah P, Singer LG, Singer JP, Sonnenday C, Tandon P, Tapper E, Tullius SG, Wilson M, Zamora M, Lai JC. Report from the American Society of Transplantation on frailty in solid organ transplantation. Am J Transplant. 2019 Apr;19(4):984-994. doi: 10.1111/ajt.15198. Epub 2018 Dec 22. PMID 30506632
- [Result] Cesari M, Marzetti E, Thiem U, Perez-Zepeda MU, Abellan Van Kan G, Landi F, Petrovic M, Cherubini A, Bernabei R. The geriatric management of frailty as paradigm of "The end of the disease era". Eur J Intern Med. 2016 Jun;31:11-4. doi: 10.1016/j.ejim.2016.03.005. Epub 2016 Mar 18. PMID 26997416
- [Result] Stuck AE, Siu AL, Wieland GD, Adams J, Rubenstein LZ. Comprehensive geriatric assessment: a meta-analysis of controlled trials. Lancet. 1993 Oct 23;342(8878):1032-6. doi: 10.1016/0140-6736(93)92884-v. PMID 8105269
- [Result] Haugen CE, Chu NM, Ying H, Warsame F, Holscher CM, Desai NM, Jones MR, Norman SP, Brennan DC, Garonzik-Wang J, Walston JD, Bingaman AW, Segev DL, McAdams-DeMarco M. Frailty and Access to Kidney Transplantation. Clin J Am Soc Nephrol. 2019 Apr 5;14(4):576-582. doi: 10.2215/CJN.12921118. Epub 2019 Mar 19. PMID 30890577
- [Result] Turner G, Clegg A; British Geriatrics Society; Age UK; Royal College of General Practioners. Best practice guidelines for the management of frailty: a British Geriatrics Society, Age UK and Royal College of General Practitioners report. Age Ageing. 2014 Nov;43(6):744-7. doi: 10.1093/ageing/afu138. PMID 25336440